CLINICAL TRIAL: NCT04655157
Title: A Multi-Center Phase I/II Open Label Study to Evaluate Safety and Efficacy in Participants With Metastatic BRAF-mutant Melanoma Treated With Encorafenib With and Without Binimetinib in Combination With Nivolumab and Low-dose Ipilimumab. (QUAD 01: Quadruple Therapy in Melanoma)
Brief Title: Safety and Efficacy in Participants With Metastatic BRAF-mutant Melanoma Treated With Encorafenib With and Without Binimetinib in Combination With Nivolumab and Low-dose Ipilimuma
Acronym: QUAD01
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated due to slow enrollment
Sponsor: Jason J. Luke, MD (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Jason J. Luke, MD, Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC 20-190; CA209-7Y4 (Other: BMS)
Record Dates: First submitted 2020-12-03; First posted 2020-12-07 (Actual); Results first posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-04

CONDITIONS: Melanoma
Keywords: BRAFV600E/K mutation; metastatic melanoma
MeSH Terms: conditions — Melanoma | interventions — encorafenib; Nivolumab; Ipilimumab; binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1 (cohort 1): 300mg encorafenib + 3mg/kg nivolumab + 1 mg/kg ipilimumab (Experimental): Patients will be treated with 300mg encorafenib and 3mg/kg nivolumab and 1 mg/kg ipilimumab (triple therapy).
  Interventions: Drug: encorafenib; Drug: nivolumab; Drug: ipilimumab
- Phase 1 (cohort 2): 450mg encorafenib + 45mg binimetinib + 3mg/kg nivolumab + 1mg/kg ipilimumab (Experimental): Patients will be treated with 450mg encorafenib, 45mg binimetinib, 3mg/kg nivolumab and 1mg/kg ipilimumab (quadruple therapy).
  Interventions: Drug: encorafenib; Drug: nivolumab; Drug: ipilimumab; Drug: binimetinib

INTERVENTIONS:
Drug: encorafenib — A small molecule BRAF inhibitor that targets key enzymes in the MAPK signaling pathway.
  Other Names: BRAFTOVI®
Drug: nivolumab — A programmed death receptor-1 (PD-1) blocking monoclonal antibody that works by helping the immune system to slow or stop the growth of cancer cells.
  Other Names: OPDIVO®
Drug: ipilimumab — A monoclonal antibody medication that works to activate the immune system by targeting CTLA-4, a protein receptor that downregulates the immune system.
  Other Names: Yervoy®
Drug: binimetinib — A small molecule, selective inhibitor of MEK, a central kinase in the tumor-promoting MAPK pathway that may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.
  Other Names: Mektovi; ARRY-162
  Arms: Phase 1 (cohort 2): 450mg encorafenib + 45mg binimetinib + 3mg/kg nivolumab + 1mg/kg ipilimumab

SUMMARY:
Patients with unresectable or metastatic BRAF-mutant melanoma high-risk patients will be given 450 mg orally (PO) daily (QD) plus binimetinib 45 mg PO twice daily (BID) together with nivolumab administered intravenously (IV) at 3mg/kg and ipilimumab administered IV at 1 mg/kg every 3 weeks for 4 doses, followed by nivolumab administered IV at 480mg every 4 weeks until progression or discontinuation due to toxicity. Concurrently, a triple therapy arm will be explored with encorafenib 300 mg PO QD together with ipilimumab administered IV at 1mg/kg and nivolumab 3mg/kg IV every 3 weeks for 4 doses, followed by nivolumab administered at 480mg every 4 weeks until progression or discontinuation due to toxicity. Tolerability of the two arms will be compared, and a recommended phase 2 dose (RP2D) will be determined. After determination of treatment schedule, expansion cohorts will further explore the preliminary efficacy and further describe the toxicity profile of the triplet or quadruplet regimen in high-risk cohorts including symptomatic brain metastases or liver metastases with elevated lactate dehydrogenase (LDH) or bulky systemic disease burden.

DETAILED DESCRIPTION:
Study participants will consist of metastatic melanoma patients harboring BRAFV600E/K mutation without previous frontline therapy or recently started treatment with up to 6 weeks of targeted therapy (or > 6 months from adjuvant therapy). Toxicity from prior treatment must have resolved to ≤ Grade 1 and not included previous Grade 3-4 immune-related adverse events (irAEs) that required treatment discontinuation or previous Grade 2 immune-related uveitis or pneumonitis.

Phase I, Cohort 1: Twelve patients will be treated with 300mg encorafenib and 3mg/kg nivolumab and 1 mg/kg ipilimumab. The dose limiting toxicity (DLT) for cohort 1 will be evaluated between weeks 1-6.

Phase I, Cohort 2: Upfront quadruple therapy with 450mg encorafenib, 45mg binimetinib, 3mg/kg nivolumab and 1mg/kg ipilimumab will be investigated with 12 participants. DLT window for phase I, cohort 2 will be evaluated at weeks 1-6.

Upon establishment of RP2R schedule, only participants with advanced melanoma who are treatment naïve in metastatic setting or have had up to 6 weeks of targeted therapy or who have progressed on adjuvant therapy for more than 6 months following completion of adjuvant therapy (either BRAF-MEK or PD1 Ab) will be eligible for participation in high risk disease cohort expansion (Groups 1 or 2).

Phase II will employ the RP2D schedule from Phase I and investigate the early efficacy in participants with high risk features who are less likely to derive benefit from standard treatment approaches and who may benefit from quadruple therapy despite the potential for increased toxicity. These will include: Group 1) symptomatic brain metastases [up to 30 patients] and Group 2) Elevated LDH >1x upper limit of normal (ULN) with: a) liver metastases OR b) bulky visceral disease (sum of longest diameter (SLD) > 44mm) [combined with Group 1 up to 60 total patients].

Following initiation of triple or quadruple therapy, participants will be followed for safety and response. Safety assessments will be a high priority with on-going Bayesian toxicity monitoring and efficacy assessments every 12 weeks. Based on prior targeted, immune, and triplet therapy studies, we anticipate up to 30-50% DLT and will consider temporary suspension of trial enrollment with a DLT > 75% as determined by CTCAEv5. Treatment efficacy will be documented using RECIST 1.1 and RANO-BM criteria, recorded every 4-12 weeks, and immune-RECIST (iRECIST) and immune-RANO (iRANO) criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent

   1. Participants must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol-related procedures that are not part of normal subject care.
   2. Participants must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study.
2. Age ≥18 years
3. Histologically confirmed diagnosis of unresectable or metastatic melanoma
4. Presence of BRAFV600E/K mutation in tumor tissue as determined in a CLIA certified laboratory
5. Patients are required to submit archival biopsy material, if available, and submit research blood samples prior to first dose. Ten patients in each Phase Ib cohort will undergo fresh biopsy. These will be the first 10 unless medical or societal factors (e.g. COVID19) limit the pursuit of research biopsies.
6. Patients must be greater than 6 months from completion of adjuvant therapy (if any given) and/or treatment naïve in the metastatic setting or have recently started targeted therapy within the last 6 weeks.
7. Prior radiotherapy must have been completed at least 2 weeks prior to study drug administration.
8. An ECOG Performance Status of 0 or 1. If enrolling in Group 1 of Phase II, can have Performance Status from 0-2.
9. Measurable disease by CT or MRI per RANO-BM (brain metastases) OR RECIST v1.1 criteria
10. Must have high risk features described as described in Phase II expansion cohort - EITHER brain metastases as described in Phase II Group 1 OR Elevated LDH/Bulky Visceral Disease as described in Phase II Group 2.
11. Adequate bone marrow, organ function, and laboratory parameters:

    1. ANC > 1.5 x 109 ¬ /L;
    2. Hemoglobin > 8 g/dL with or without transfusions;
    3. Platelet > 100 x 109 ¬ /L;
    4. Serum creatinine ≤ 1.5 × ULN, OR calculated creatinine clearance > 50 mL/min by Cockcroft-Gault formula, OR estimated glomerular filtration rate > 50 mL/min/1.73 m
12. Patient IS permitted to be on corticosteroids if related to disease burden and MAY have symptomatic brain lesions as long as radiation or surgical intervention is not deemed to be urgently necessary.

    1. Symptomatic intracranial metastases may be on steroids at a total daily dose of no higher than 4 mg of dexamethasone or equivalent that is stable or tapering for 10 days prior to first treatment,
    2. have no immediate need for SRT or surgery (within 3 week prior to first treatment),
    3. have a performance status of 0-2 and
    4. have had no experience of seizure within 10 days prior to first treatment.
13. Female patients of childbearing potential must have a negative serum β-HCG test result during screening prior to first dose
14. Females of childbearing potential must agree to protocol-approved methods of contraception, and to not donate Ova from Screening until 30 days of last dose of study drug.
15. Male patients must use contraception that is highly effective or acceptable, and not donate sperm from Screening until 90 days after the last dose of study drug.
16. The patient is deemed by the Investigator to have the initiative and means to comply with scheduled visits, treatment plan and study procedures.

Exclusion Criteria:

1. Known hypersensitivity or contraindication to any component of study treatment or their excipients.
2. Previous Grade 3-4 AEs, or discontinuation of PD-1 or CTLA-4 inhibitor therapy, or BRAF/MEK inhibitor therapy
3. Inability to swallow and retain study treatment
4. Impairment of gastrointestinal function or disease which may significantly alter the absorption of study treatment (e.g., active ulcerative disease; uncontrolled nausea, vomiting or diarrhea; malabsorption syndrome; small bowel resection).
5. Participants with a non-melanoma related condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
6. Participants with active, known or suspected autoimmune disease including those who have required systemic anti-rheumatic therapies in the preceding 2 years. Participants with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
7. Impaired cardiovascular function or clinically significant cardiovascular disease including, but not limited to, the following:

   1. History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty or stenting) < 6 months prior to Screening
   2. Congestive heart failure requiring treatment (New York Heart Association Grade ≥ 2)
   3. A known LVEF < 50% as determined by MUGA or ECHO
   4. Uncontrolled hypertension defined as persistent systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg despite current therapy
   5. History or presence of clinically significant cardiac arrhythmias (including resting bradycardia, uncontrolled atrial fibrillation or uncontrolled paroxysmal supraventricular tachycardia)
   6. Baseline QTcF interval ≥ 480 ms.
8. Second malignancy that requires active treatment or would interfere with treatment efficacy evaluation. Participants with a second malignancy treated with curative intent are eligible.
9. On-going or use of systemic antibiotics during the preceding 2 weeks prior to enrollment
10. Known acute or chronic infection with hepatitis B or hepatitis C virus. Participants treated with curative anti-viral therapy are eligible.
11. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) even if fully immunocompetent on ART-due to the unknown effects of HIV on the immune response to combined nivolumab plus ipilimumab or the unique toxicity spectrum of these drugs in patients with HIV.
12. History of a thromboembolic event < 12 weeks prior to starting study treatment. Examples of thromboembolic events include transient ischemia attack, cerebrovascular accident, deep vein thrombosis or pulmonary embolism. Catheter-related venous thrombosis is not considered a thromboembolic event for this trial even if < 12 weeks prior to starting study treatment.
13. Use of herbal supplements, medications or foods that are moderate or strong inhibitors or inducers of cytochrome P450 (CYP) 3A4/5 ≤ 1 week prior to the start of study treatment (Section 4.5.1).
14. History or current evidence of RVO or current risk factors for RVO (e.g., uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes); history of retinal degenerative disease.

Phase II Group 1 Specific Criteria

1. For Phase II Group 1 (Brain Metastases): Patients may have an ECOG status of 0-2 and IS permitted to be on corticosteroids if related to disease burden and MAY have symptomatic brain lesions as long as radiation or surgical intervention is not deemed to be urgently necessary.

1. Symptomatic intracranial metastases may be on steroids at a total daily dose of no higher than 4 mg of dexamethasone or equivalent that is stable or tapering for 10 days prior to first treatment,
2. have no immediate need for SRT or surgery (within 3 week prior to first treatment),
3. have had no experience of seizure within 10 days prior to first treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason J Luke, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phase 1 (Cohort 1): 300mg Encorafenib + 3mg/kg Nivolumab + 1 mg/kg Ipilimumab | Phase 1 (Cohort 2): 450mg Encorafenib + 45mg Binimetinib + 3mg/kg Nivolumab + 1mg/kg Ipilimumab
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 (Cohort 1): 300mg Encorafenib + 3mg/kg Nivolumab + 1 mg/kg Ipilimumab | Phase 1 (Cohort 2): 450mg Encorafenib + 45mg Binimetinib + 3mg/kg Nivolumab + 1mg/kg Ipilimumab | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 32 [32 to 32] | 65 [65 to 65] | 48.5 [32 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase II Dose (RP2D) of Encorafenib + Nivolumab + Ipilimumab
Description: Determination of recommended phase II dose (RP2D) of triple therapy in patients treated with 300mg encorafenib, 3mg/kg nivolumab and 1mg/kg ipilimumab via the frequency of DLTs that are classified as either possibly, probably, or definitely related to study treatment according to NCI Common Terminology Criteria for Adverse Events (CTCAE v5.0). Number of distinct patients experiencing Adverse events and DLTs. This will be done with continuous Bayesian toxicity monitoring.
Time Frame: Up to 6 weeks (DLT evaluation period)
Population: Patients that received treatment
Measure: Number; unit: mg
Arm/Group | Phase 1 (Cohort 1): 300mg Encorafenib + 3mg/kg Nivolumab + 1 mg/kg Ipilimumab
Number analyzed (Participants) | 1
mg | NA — RP2D cannot be determined due to insufficient number of participants

2. Primary Outcome: Recommended Phase II Dose (RP2D) of Encorafenib + Binimetinib + Nivolumab + Ipilimumab
Description: Determination of recommended phase II dose (RP2D) of quadruple therapy in patients treated with 450mg encorafenib, 45mg binimetinib, 3mg/kg nivolumab and 1mg/kg ipilimumab via the frequency of DLTs that are classified as either possibly, probably, or definitely related to study treatment according to NCI Common Terminology Criteria for Adverse Events (CTCAE v5.0). Number of distinct patients experiencing Adverse events and DLTs. This will be done with continuous Bayesian toxicity monitoring.
Time Frame: Up to 6 weeks (DLT evaluation period)
Population: Patients that received treatment
Measure: Number; unit: mg
Groups:
- Phase 1 (Cohort 2): 450 mg Encorafenib + 45mg Binimetinib + 3mg/kg Nivolumab + 1mg/kg Ipilimumab: Patients will be treated with 450 mg encorafenib, 45mg binimetinib, 3mg/kg nivolumab and 1mg/kg ipilimumab (quadruple therapy).
  encorafenib: A small molecule BRAF inhibitor that targets key enzymes in the MAPK signaling pathway.
  nivolumab: A programmed death receptor-1 (PD-1) blocking monoclonal antibody that works by helping the immune system to slow or stop the growth of cancer cells.
  ipilimumab: A monoclonal antibody medication that works to activate the immune system by targeting CTLA-4, a protein receptor that downregulates the immune system.
  binimetinib: A small molecule, selective inhibitor of MEK, a central kinase in the tumor-promoting MAPK pathway that may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.
Arm/Group | Phase 1 (Cohort 2): 450 mg Encorafenib + 45mg Binimetinib + 3mg/kg Nivolumab + 1mg/kg Ipilimumab
Number analyzed (Participants) | 1
mg | NA — RP2D cannot be determined due to insufficient number of participants

3. Secondary Outcome: Response Rate Per RECIST v1.1 Criteria
Description: Number of patients with Complete response [CR] + partial response [PR], per RECIST v1.1 criteria . Per RECIST v1.1, CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. For non-target lesions: Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10mm short axis); PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 15 months
Population: Patients receiving at least one dose any drug and/or evaluable for response
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 (Cohort 1): 300mg Encorafenib + 3mg/kg Nivolumab + 1 mg/kg Ipilimumab | Phase 1 (Cohort 2): 450mg Encorafenib + 45mg Binimetinib + 3mg/kg Nivolumab + 1mg/kg Ipilimumab
Number analyzed (Participants) | 1 | 1
Participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 0 | 0

4. Secondary Outcome: Central Nervous System (CNS) Clinical Benefit Rate (CBR)
Description: Number of patients with Complete response [CR] + partial response [PR] + stable disease [SD] >6 months) per RANO-BM criteria. Per RANO, CR: No lesion present; PR: ≥30% decrease in sum LD relative to baseline; SD: <30% decrease relative to baseline, but <20% increase in sum LD relative to nadir.
Time Frame: Up to 15 months
Population: Patients receiving at least one dose any drug and/or evaluable for response
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 (Cohort 1): 300mg Encorafenib + 3mg/kg Nivolumab + 1 mg/kg Ipilimumab | Phase 1 (Cohort 2): 450mg Encorafenib + 45mg Binimetinib + 3mg/kg Nivolumab + 1mg/kg Ipilimumab
Number analyzed (Participants) | 1 | 1
Participants
  Complete Response | 0 | 0
  Partial Reponse | 0 | 0
  Stable Disease | 1 | 0

5. Secondary Outcome: Adverse Events at Least Probably Related to Treatment
Description: Number of (distinct) participants with ≤ Grade 3 Adverse Events or Serious Adverse Events that are possibly, probably or definitely related to study treatment per the Criteria for Adverse Events version 5 (CTCAEv5).
Time Frame: Up to 6 months (per patient)
Population: Patients receiving at least one dose of (any) study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 (Cohort 1): 300mg Encorafenib + 3mg/kg Nivolumab + 1 mg/kg Ipilimumab | Phase 1 (Cohort 2): 450mg Encorafenib + 45mg Binimetinib + 3mg/kg Nivolumab + 1mg/kg Ipilimumab
Number analyzed (Participants) | 1 | 1
Participants
  Arthralgia | 1 | 0
  Myalgia | 1 | 0
  Fever | 1 | 0
  Hypotension | 1 | 0
  Anemia | 1 | 0
  ALT Increased | 1 | 0
  Dyspnea | 1 | 0
  Hypokalemia | 1 | 0
  Hypertension | 1 | 0
  Lymphocyte decreased | 1 | 0

6. Secondary Outcome: Progression-free Survival (PFS)
Description: The length of time during and after study treatment that each patient lived with cancer but it does not get worse. PFS is one way to assess how the treatment works. Per RECIST v1.1, progressive disease is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. For non-target lesions, PD: Unequivocal progression of existing non-target lesions. The appearance of one or more new lesions is also considered progression.
Time Frame: Up to 15 months
Population: Includes patients receiving at least one dose any drug and/or evaluable for response
Measure: Number; unit: months
Arm/Group | Phase 1 (Cohort 1): 300mg Encorafenib + 3mg/kg Nivolumab + 1 mg/kg Ipilimumab | Phase 1 (Cohort 2): 450mg Encorafenib + 45mg Binimetinib + 3mg/kg Nivolumab + 1mg/kg Ipilimumab
Number analyzed (Participants) | 1 | 1
months | 6 | 3

ADVERSE EVENTS:
Time Frame: Adverse Events data were collected for up to 6 months per patient and up to 15 months overall duration for study.
Arm/Group | Phase 1 (Cohort 1): 300mg Encorafenib + 3mg/kg Nivolumab + 1 mg/kg Ipilimumab | Phase 1 (Cohort 2): 450mg Encorafenib + 45mg Binimetinib + 3mg/kg Nivolumab + 1mg/kg Ipilimumab
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1 | 1/1
Other Adverse Events (participants affected / at risk) | 1/1 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 (Cohort 1): 300mg Encorafenib + 3mg/kg Nivolumab + 1 mg/kg Ipilimumab (N=1) | Phase 1 (Cohort 2): 450mg Encorafenib + 45mg Binimetinib + 3mg/kg Nivolumab + 1mg/kg Ipilimumab (N=1)
Spinal Cord Compression (Nervous system disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 — inflammation and thoracic/lumbar spinal disease
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 (Cohort 1): 300mg Encorafenib + 3mg/kg Nivolumab + 1 mg/kg Ipilimumab (N=1) | Phase 1 (Cohort 2): 450mg Encorafenib + 45mg Binimetinib + 3mg/kg Nivolumab + 1mg/kg Ipilimumab (N=1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
ALT Increased (Investigations) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Lymphocyte decreased (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT04655157/Prot_SAP_000.pdf